CLINICAL TRIAL: NCT02331589
Title: Anti-fatigue Effect of Korean Red Ginseng in Patients With Non-alcoholic Hepatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Ki Tae Suk, doctor, assistant professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFEKRG
Record Dates: First submitted 2014-12-31; First posted 2015-01-06 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2014-12

CONDITIONS: Fatigue
Keywords: Fatigue; Panax ginseng; Chronic hepatitis; Non-alcoholic Fatty Liver Disease; Adiponectin
MeSH Terms: conditions — Fatigue; Hepatitis, Chronic; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Korea Red Ginseng (KRG) (Active Comparator): KRG capsule (3,000 mg/day) for 3 weeks
  Interventions: Drug: KRG (Korea Red ginseng)
- Placebo (for KRG) (Placebo Comparator): placebo (for KRG) for 3 weeks
  Interventions: Drug: Placebo (for KRG)

INTERVENTIONS:
Drug: KRG (Korea Red ginseng) — 3 weeks of KRG capsule (3,000 mg/day)
  Other Names: Korea Red ginseng capsule (3,000 mg/day)
  Arms: Korea Red Ginseng (KRG)
Drug: Placebo (for KRG) — Placebos with same shape and size were manufactured and at Korea Ginseng Corporation
  Other Names: Placebo
  Arms: Placebo (for KRG)

SUMMARY:
Background: Korea red ginseng (KRG) has anti-carcinogenic activity, anti-oxidant activity, and cancer related anti-fatigue.

Methods: Seventy five patients with non-alcoholic hepatitis were prospectively randomized to receive 3 weeks of KRG or placebo. Liver function test, pro-inflammatory cytokines, adiponectin, fatigue severity scale, and antioxidant activity were check and compared.

DETAILED DESCRIPTION:
Fatigue Severity Scale

We used to be KRUPP's fatigue severity scale. The survey has nine questions as following: (1) my motivation is lower, when I am fatigued (2) exercise brings on my fatigue (3) I am easily fatigued (4) fatigue interferes with my physical functioning (5) fatigue causes frequent problems for me (6) my fatigue prevents sustained physical functioning (7) fatigue interferes with carrying out certain duties and responsibilities (8) fatigue is among my 3 most disabling symptoms (9) fatigue interferes with my work, family, or social life. All subjects scored each question on a 7-point scale (1 = strongly disagree to 4 = neither disagree nor agree to 7 = strongly agree). All fatigue severity scale calculated and collected by one research nurse (C.W.K) in the Department of Internal Medicine.

ELIGIBILITY:
Inclusion Criteria:

* aspartate aminotransferase (AST) ≥ 50 U/L or alanine aminotransferase (ALT) ≥ 50 U/L, and Fatty liver or Hepatitis

Exclusion Criteria:

* viral hepatitis, alcoholic hepatitis, autoimmune hepatitis, pancreatitis, hemochromatosis, Wilson's disease, drug induced liver injury, or cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Korea Red Ginseng (KRG) | Placebo (for KRG)
Started | 39 | 36
Completed | 34 | 31
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Korea Red Ginseng (KRG) | Placebo (for KRG) | Total
Number analyzed (Participants) | 34 | 31 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 27 | 58
  >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (12.7) | 50.0 (12.8) | 47.8 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 27 | 26 | 53
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 34 | 31 | 65

OUTCOME MEASURES:

1. Primary Outcome: Liver Enzymes
Description: aspartate aminotransferase, alanine aminotransferase, gamma glutamyl transferase, lactate dehydrogenase
Time Frame: 3 weeks of KRG
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Korea Red Ginseng (KRG) | Placebo (for KRG)
Number analyzed (Participants) | 35 | 31
U/L
  aspartate aminotransferase | 52.1 (30.7) | 59.1 (37.2)
  alanine aminotransferase | 81.0 (43.7) | 81.6 (32.2)
  gamma glutamyl transferase | 106.9 (68.6) | 139.3 (198.2)
  lactate dehydrogenase | 226.7 (99.0) | 218.6 (34.1)

2. Secondary Outcome: Fatigue as Measured by KRUPP's Fatigue Severity Scale
Description: KRUPP's fatigue severity scale.
  The survey has nine questions as following:
  1. my motivation is lower, when I am fatigued
  2. exercise brings on my fatigue
  3. I am easily fatigued
  4. fatigue interferes with my physical functioning
  5. fatigue causes frequent problems for me
  6. my fatigue prevents sustained physical functioning
  7. fatigue interferes with carrying out certain duties and responsibilities
  8. fatigue is among my 3 most disabling symptoms
  9. fatigue interferes with my work, family, or social life. All subjects scored each question on a 7-point scale (1 = strongly disagree to 4 = neither disagree nor agree to 7 = strongly agree).
  Scores range from 9 to 63, with higher scores indicating higher fatigue
Time Frame: 3 weeks of KRG
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Korea Red Ginseng (KRG) | Placebo (for KRG)
Number analyzed (Participants) | 35 | 31
scores on a scale | 33.0 (11.6) | 29.8 (14.1)

3. Secondary Outcome: Pro-inflammatory Cytokine
Description: tumor necrosis factor-alpha, interleukin-6
Time Frame: 3 weeks of KRG
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Korea Red Ginseng (KRG) | Placebo (for KRG)
Number analyzed (Participants) | 35 | 31
pg/mL
  tumor necrosis factor-alpha | 108.0 (54.8) | 123.1 (42.1)
  interleukin-6 | 2.3 (1.9) | 1.5 (0.4)

4. Secondary Outcome: Adiponectin
Description: enzyme-linked immunosorbent assay
Time Frame: 3 weeks of KRG
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Korea Red Ginseng (KRG) | Placebo (for KRG)
Number analyzed (Participants) | 35 | 31
pg/mL | 7751.2 (3108.1) | 7711.6 (3041.3)

ADVERSE EVENTS:
Time Frame: Serious and Other (Not Including Serious) Adverse Events were not collected/assessed
Arm/Group | Korea Red Ginseng (KRG) | Placebo (for KRG)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other